CLINICAL TRIAL: NCT02984033
Title: Quality of Life and Psychological Evaluation of Patients Affected by Head and Neck Cancer Treated With Curative Intent: Multicentric Prospective Study
Brief Title: Quality of Life and Psycological Evaluation of Patients Affected by Head and Neck Cancer
Status: Withdrawn | Type: Observational
Why Stopped: No patient enrolled
Sponsor: Michele Tedeschi (Other)
Responsible Party: Sponsor-Investigator, Michele Tedeschi, Medical Doctor, Istituto Clinico Humanitas
Organization: Istituto Clinico Humanitas (Other)
Other Study IDs: 1642
Record Dates: First submitted 2016-12-02; First posted 2016-12-06 (Estimated); Last update posted 2018-10-24 (Actual); Status verified 2018-10

CONDITIONS: Quality of Life

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (1):
- Head and Neck patients: Patients affected by squamous cell carcinoma of head and neck (oral cavity, larynx, pharynx and hypopharynx) with no metastasis
  Interventions: Radiation: Head and Neck patients

INTERVENTIONS:
Radiation: Head and Neck patients — Treatment consists of Intensity Modulated Radiation Therapy (until 2.2 Gy) with a total dose of 50-66 Gy in post-operative setting and 66-72 Gy in radical setting.

SUMMARY:
The prospective trial is to describe the quality of life and psychological effects in patients with head and neck tumor receiving curative intent treatment

DETAILED DESCRIPTION:
The multicentric prospective trial is to evaluate the quality of life and psychological effects in patients with head and neck tumor treated by curative intent radiation therapy. The treatment consists in a conventionally fractionated Intensity Modulated Radiotherapy (IMRT) or until 2.2 Gy per fraction with a total dose of 50-66 Gy in post-operative setting and 66-72 Gy in radical setting.

ELIGIBILITY:
Inclusion Criteria:

* Squamous cell carcinoma of head and neck (oral cavity, larynx, pharynx and hypopharynx) in non-metastatic staging;
* curative intent treatment (radiation therapy associated or not to chemotherapy; surgery associated or not to post-operative radiotherapy and chemotherapy);
* performance status < 2;
* age ≥ 18 years;
* good knowledge of italian language;
* written informed consent

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients affected by head and neck tumor
Sampling Method: Non-Probability Sample
Enrollment: 0 (Actual)
Dates: Start 2016-11; Primary Completion 2018-02-01 (Actual); Study Completion 2018-02-01 (Actual)

PRIMARY OUTCOMES:
Quality of life and psychological effetcs evaluated by patient reported outcome (PRO) | 18 months

CONTACTS AND LOCATIONS:
Overall Officials: Ciro Franzese, MD, Study Chair — Humanitas Cancer Center
Locations (1):
- Humanitas Research Hospital, Rozzano, Milano, Italy

IPD SHARING:
Plan to Share IPD: No